CLINICAL TRIAL: NCT04532164
Title: HT201309- Human Photoallergy Test
Brief Title: Study to Find Out if Cream V61-044 Used to Treat Fungal Infections Causes an Allergic Skin Reaction to Sunlight in Healthy Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18155
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Dermatitis, Photoallergic
MeSH Terms: conditions — Dermatitis, Photoallergic | interventions — butenafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Photoallergic reaction test (Experimental): During the Induction Phase, participants received Butenafine HCl 1% on the treated irradiated skin test site followed by UV irradiation and on the treated non-irradiated skin test site without UV radiation, two times per week for three consecutive weeks. After 10 days of Rest Phase, during the Challenge Phase, participants received same procedure on the two virgin sites (treated sites) as in Induction Phase, and two additional sites with no Butenafine HCl 1% (untreated sites) were also occluded. Test sites were evaluated at 24, 48, and 72 hours after irradiation using the same grading scale used during Induction Phase.
  Interventions: Drug: Butenafine HCl 1% (BAY1896425) - Induction Phase; Drug: Butenafine HCl 1% (BAY1896425) - Challenge Phase

INTERVENTIONS:
Drug: Butenafine HCl 1% (BAY1896425) - Induction Phase — To each of two test sites, approximately 20 μl/cm^2 of the Butenafine HCl 1% was applied directly to the skin and covered with a 25 mm Hilltop chamber with a Webril pad (2 cm in diameter, within an area of approximately 3 cm^2), and tape was applied over the chamber to secure the occlusive patch to the skin. On the next day, the chambers were removed and both test sites were lightly wiped. Approximately 2 μl/cm^2 of Butenafine HCl 1% was reapplied directly to the skin and lightly spread over the treated irradiated test site. The treated non-irradiated test site did not receive a similar reapplication. Between 5 and 15 minutes after application, the treated irradiated test site was irradiated with two times the subject's Minimal Erythema Dose (MED). Evaluation of the test sites occurred two days after the irradiation. This procedure was repeated two times per week for three consecutive weeks for a total of 6 induction exposures per test site.
  Other Names: Antifungal Cream V61-044 containing Trolamine
Drug: Butenafine HCl 1% (BAY1896425) - Challenge Phase — 5 μl/cm^2 of the Butenafine HCl 1% was applied directly to each of the two virgin sites (treated sites) adjacent to the induction patch sites and covered with Hilltop chambers with Webril pad and tape was applied over the chambers to secure the occlusive patches to the skin. Two additional sites with no Butenafine HCl 1% (untreated sites) were also occluded. Sites were at least 2.5 cm apart. The patches were removed 24 hours later and the sites were lightly wiped. Test sites were evaluated. Butenafine HCl 1% (2 μl/cm^2) was applied to the treated irradiated site. After 15 minutes, the treated irradiated site and the untreated irradiated site were irradiated with 0.5 MED of UVA/UVB irradiation followed by 10 Joules/cm^2 of UVA from a xenon arc solar simulator equipped with a Schott WG345 to eliminate UVB radiation. The remaining sites served as the treated non-irradiated site and untreated non-irradiated site.
  Other Names: Antifungal Cream V61-044 containing Trolamine

SUMMARY:
Allergic skin reaction can be produced by the combination of a chemical product applied to the skin and ultraviolet (UV) radiation (a type of invisible light that comes from the sun and other light sources and can hurt your skin and eyes) received by the person. The researchers in this study wanted to find out if cream V61-044 might cause an allergic skin reaction to sunlight when applied to the skin in healthy participants. Cream V61-044 (brand name: LOTRIMIN ULTRA) is an approved drug used to treat infections caused by fungi (small growing organisms such as mold, mildew, yeast or mushrooms).

Participants joining this study underwent two study phases: in Induction phase, participants received the test cream and UV radiation twice a week for 3 weeks; after 10 days of rest, in Challenge phase participants received the test cream and UV radiation once again. In both phases, the test cream was applied to two test areas on the upper back of the participants and to one of the test area UV radiation was applied. Evaluation on the skin rash was conducted two days after each UV radiation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been between the ages of 18 and 60 years;
* Subjects must have been lightly pigmented with skin phototypes I - III, determined by the following guidelines: I-Always burns easily; never tans (sensitive); II-Always burns easily; tans minimally (sensitive); III-Burns moderately; tans gradually (light-brown) (normal);
* Subjects must have been in general good health as determined by the subject's medical history;
* Subjects must have been willing to avoid tanning bed usage and additional sun exposure during the study and follow-up period;
* Subjects must have been willing to refrain from using any new topical products during the trial;
* Subjects must have been able and willing to cooperate with the Investigator and research staff, to have test materials applied according to protocol, and to complete the full course of the trial;
* Subjects must have been willing to report any medications taken during the trial and refrain from taking any medications during the trial that might produce photoreactions;
* If female, produced a negative urine pregnancy test prior to the initiation and also at the completion of the study.

Exclusion Criteria:

* Subjects with a visible sunburn;
* Subjects who had a history of sun hypersensitivity, photosensitivity, or photosensitive dermatoses;
* Subjects with a history of allergies or sensitivities to cosmetics, toiletries, or any dermatological products;
* Subjects who had recently used any systemic or topical drugs which can cause a photoreaction or may interfere with the trial;
* Subjects with any known skin conditions that might have interfered with the proper conduct of the trial;
* Subjects with scars, moles, excessive hair, or other blemishes over the mid or lower back which might have interfered with the test or the grading of the test sites;
* Subjects who had significant history of internal disease that may have interfered with the evaluation of the test material as determined by the Investigator;
* Female subjects who were pregnant, planning pregnancy, or nursing a child during the study period;
* Subjects who had used a tanning bed or other artificial tanning lights within the past two months;
* Subjects who had participated in a patch test involving the back within four weeks prior to the start of the trial;
* Subjects who would concurrently participate in any other clinical or consumer test;
* Subjects who had other conditions considered by the Investigator as sound reasons for disqualification from enrollment into the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2013-11-11 (Actual); Study Completion 2013-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at single center in the US, between 10 JUN 2013 (first subject first visit) and 11 NOV 2013 (last subject last visit).
Pre-assignment Details: A total of 137 subjects were enrolled in the study and 132 received study treatment.
Period: Overall Study
Arm/Group | Photoallergic Reaction Test
Started | 137
Treated | 132
Completed | 113
Not Completed | 24
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 1
Not completed — Found to be Ineligible | 3
Not completed — Withdrawal by Subject | 14

BASELINE CHARACTERISTICS:
Arm/Group | Photoallergic Reaction Test
Number analyzed (Participants) | 137
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 48
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 99
  Hispanic | 34
  Caucasian/Hispanic | 2
  Asian | 1
  Caucasian/Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Photoallergic Reaction Evaluation Reported as Number of Test Site With Different Erythema Score During Challenge Phase - All Treated Subjects
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=normal skin (no visible reaction); score 1= faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=moderate to intense redness with well defined margins; score 3=redness with well defined edema; score 4=redness with papules, vesicles, or ulceration. During Challenge Phase, each subject had the following four virgin test sites: Treated irradiated test site; Treated non-irradiated test site; Untreated irradiated test site; Untreated non-irradiated test site. All four test sites were evaluated according to the above scoring system at 24, 48, and 72 hours following patch application (3 different time points), and the number of test sites with available scores from all these time points were reported for all treated subjects.
Time Frame: At 24, 48, and 72 hours following patch application
Population: Subjects who received treatment
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Challenge Phase
Number analyzed (Participants) | 132
Number analyzed (Test site) | 349
Test site
  Treated irradiated test site, score=0 | 325
  Treated irradiated test site, score=1 | 24
  Treated non-irradiated test site, score=0 | 343
  Treated non-irradiated test site, score=1 | 6

2. Secondary Outcome: Development of Erythema on Treated Irradiated Test Sites During Induction Phase - All Treated Subjects
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=normal skin (no visible reaction); score 1= faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=moderate to intense redness with well defined margins; score 3=redness with well defined edema; score 4=redness with papules, vesicles, or ulceration. During Induction Phase, each subject had the following two test sites: Treated irradiated test site and Treated non-irradiated test site. The number of test sites with available scores from all 6 induction patches were reported for all treated subjects.
Time Frame: Two or three days after each irradiation during Induction Phase
Population: Subjects who received treatment
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Groups:
- Butenafine HCl 1% (BAY1896425) - Induction Phase: To each of two test sites, approximately 20 μl/cm^2 of the Butenafine HCl 1% was applied directly to the skin and covered with a 25 mm Hilltop chamber with a Webril® pad (2 cm in diameter, within an area of approximately 3 cm^2), and tape was applied over the chamber to secure the occlusive patch to the skin. On the next day, the chambers were removed and both test sites were lightly wiped. Approximately 2 μl/cm^2 of Butenafine HCl 1% was reapplied directly to the skin and lightly spread over the treated irradiated test site. The treated non-irradiated test site did not receive a similar reapplication. Between 5 and 15 minutes after application, the treated irradiated test site was irradiated with two times the subject's Minimal Erythema Dose (MED). Evaluation of the test sites occurred two days after the irradiation. This procedure was repeated two times per week for three consecutive weeks for a total of 6 induction exposures per test site.
Arm/Group | Butenafine HCl 1% (BAY1896425) - Induction Phase
Number analyzed (Participants) | 132
Number analyzed (Test site) | 630
Test site
  Treated irradiated test site, score=0 | 273
  Treated irradiated test site, score=1 | 282
  Treated irradiated test site, score=2 | 75

3. Secondary Outcome: Development of Erythema on the Treated Non-irradiated Test Sites During Induction Phase - All Treated Subjects
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=normal skin (no visible reaction); score 1= faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=moderate to intense redness with well defined margins; score 3=redness with well defined edema; score 4=redness with papules, vesicles, or ulceration. During Induction Phase, each subject had the following two test sites: Treated irradiated test site and Treated non-irradiated test site. The mean score of test sites with available scores from all 6 induction patches were reported for all treated subjects.
Time Frame: Two or three days after each irradiation during Induction Phase
Population: Subjects who received treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Induction Phase
Number analyzed (Participants) | 132
Number analyzed (Test site) | 630
Score on a scale | 0 (0)

4. Secondary Outcome: Development of Erythema on the Treated Non-irradiated Test Sites During Challenge Phase Reported as Number of Test Site With Different Erythema Score - All Treated Subjects
Description: as for outcome 1
Time Frame: At 24, 48, and 72 hours following patch application
Population: Subjects who received treatment
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Challenge Phase
Number analyzed (Participants) | 132
Number analyzed (Test site) | 349
Test site
  Treated non-irradiated test site, score=0 | 343
  Treated non-irradiated test site, score=1 | 6

5. Primary Outcome: Photoallergic Reaction Evaluation Reported as Number of Test Site With Different Erythema Score During Challenge Phase - All Evaluable Subjects
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=normal skin (no visible reaction); score 1= faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=moderate to intense redness with well defined margins; score 3=redness with well defined edema; score 4=redness with papules, vesicles, or ulceration. During Challenge Phase, each subject had the following four virgin test sites: Treated irradiated test site; Treated non-irradiated test site; Untreated irradiated test site; Untreated non-irradiated test site. All four test sites were evaluated according to the above scoring system at 24, 48, and 72 hours following patch application (3 different time points), and the number of test sites with available scores from all these time points were reported for all evaluable subjects.
Time Frame: At 24, 48, and 72 hours following patch application
Population: Subjects who received treatment and completed the trial and had evaluable data
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Challenge Phase
Number analyzed (Participants) | 107
Number analyzed (Test site) | 320
Test site
  Treated irradiated test site, score=0 | 311
  Treated irradiated test site, score=1 | 9
  Treated non-irradiated test site, score=0 | 314
  Treated non-irradiated test site, score=1 | 6

6. Secondary Outcome: Development of Erythema on Treated Irradiated Test Sites During Induction Phase - All Evaluable Subjects
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=normal skin (no visible reaction); score 1= faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=moderate to intense redness with well defined margins; score 3=redness with well defined edema; score 4=redness with papules, vesicles, or ulceration. During Induction Phase, each subject had the following two test sites: Treated irradiated test site and Treated non-irradiated test site. The number of test sites with available scores from all 6 induction patches were reported for all evaluable subjects.
Time Frame: Two or three days after each irradiation during Induction Phase
Population: Subjects who received treatment and completed the trial and had evaluable data
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Induction Phase
Number analyzed (Participants) | 107
Number analyzed (Test site) | 540
Test site
  Treated irradiated test site, score=0 | 248
  Treated irradiated test site, score=1 | 231
  Treated irradiated test site, score=2 | 61

7. Secondary Outcome: Development of Erythema on the Treated Non-irradiated Test Sites During Induction Phase - All Evaluable Subjects
Description: Evaluation of the test sites after irradiation used following scoring system: score 0=normal skin (no visible reaction); score 1= faint, barely perceptible to moderate redness with poorly defined margins (not clinically significant); score 2=moderate to intense redness with well defined margins; score 3=redness with well defined edema; score 4=redness with papules, vesicles, or ulceration. During Induction Phase, each subject had the following two test sites: Treated irradiated test site and Treated non-irradiated test site. The mean score of test sites with available scores from all 6 induction patches were reported for all evaluable subjects.
Time Frame: Two or three days after each irradiation during Induction Phase
Population: Subjects who received treatment and completed the trial and had evaluable data
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Induction Phase
Number analyzed (Participants) | 107
Number analyzed (Test site) | 540
Score on a scale | 0 (0)

8. Secondary Outcome: Development of Erythema on the Treated Non-irradiated Test Sites During Challenge Phase Reported as Number of Test Site With Different Erythema Score - All Evaluable Subjects
Description: as for outcome 5
Time Frame: At 24, 48, and 72 hours following patch application
Population: Subjects who received treatment and completed the trial and had evaluable data
Measure: Number; unit: Test site
Units Other Than Participants: Test site
Arm/Group | Butenafine HCl 1% (BAY1896425) - Challenge Phase
Number analyzed (Participants) | 107
Number analyzed (Test site) | 320
Test site
  Treated non-irradiated test site, score=0 | 314
  Treated non-irradiated test site, score=1 | 6

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Photoallergic Reaction Test
Serious Adverse Events (participants affected / at risk) | 1/137
Other Adverse Events (participants affected / at risk) | 8/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photoallergic Reaction Test (N=137)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Photoallergic Reaction Test (N=137)
Toothache (Gastrointestinal disorders) | 1 (1)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Other (Ankle Sprain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Other (Insect Bite) (Infections and infestations) | 1 (1)
Eye Infection (Infections and infestations) | 1 (1)
Watery eyes (Eye disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No information based on the conduct of the study (incl. protocol, data resulting from the study, or the fact that the study was being conducted) will be released without prior written consent of the sponsor unless the requirement is superseded by State or Federal law.